CLINICAL TRIAL: NCT03423147
Title: A Randomized Trial to Determine if a Pre-operative Wash With a Chlorhexidine Gluconate Cloth and Chlorhexidine Gluconate Vaginal Scrub Reduces Infectious Morbidity in Patients Undergoing Cesarean Section After Labor
Brief Title: Preoperative Application of Chlorhexidine to Reduce Infection With Cesarean Section After Labor
Acronym: PRACTICAL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor enrollment, inability to achieve required number of subjects
Sponsor: Angela Bianco (Other)
Collaborators: Stryker Nordic (Industry)
Responsible Party: Sponsor-Investigator, Angela Bianco, Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GCO 17-1235
Record Dates: First submitted 2018-01-31; First posted 2018-02-06 (Actual); Results first posted 2023-03-23 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2022-02

CONDITIONS: Cesarean Section; Surgical Site Infection; Nosocomial Infection
Keywords: Cesarean section; Labor; Surgical Site Infections; Chlorhexidine gluconate
MeSH Terms: conditions — Surgical Wound Infection; Cross Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Chlorhexidine gluconate vaginal scrub and cloth (Experimental): Patients will have a 2% chlorhexidine gluconate cloth applied to their abdomen as well as 4% chlorhexidine gluconate vaginal scrub applied as a vaginal cleanse in the operating room prior to cesarean section
  Interventions: Drug: 2% chlorhexidine gluconate cloth; Drug: 4% Chlorhexidine gluconate vaginal scrub
- Standard Treatment (Active Comparator): Patients who are not in the intervention arm will receive the standard of care prior to a cesarean section. In the operating room the patient will receive an abdominal cleanse with 2% Chloraprep solution (2% chlorhexidine gluconate) in addition to routine IV antibiotics.
  Interventions: Drug: 2% chlorhexidine gluconate cloth

INTERVENTIONS:
Drug: 2% chlorhexidine gluconate cloth — applied to their abdomen
  Other Names: 2% Chloraprep solution
Drug: 4% Chlorhexidine gluconate vaginal scrub — applied as a vaginal cleanse in the operating room prior to cesarean section
  Arms: Chlorhexidine gluconate vaginal scrub and cloth

SUMMARY:
Surgical site infections (SSI) are the second most common cause of nosocomial infections accounting for 15% of all nosocomial infections among hospitalized patients and 38% of nosocomial infections in surgical patients. In obstetric patients, infectious morbidity (i.e. SSI, endometritis) occurs in 5-10% of cesarean sections, which is 5-fold higher than vaginal deliveries. Additionally, infectious morbidity is thought to be highest in those patients who have cesarean sections after undergoing labor.

Chlorhexidine, a chemical antiseptic effective on gram positive and gram negative bacteria, reduces skin microflora/colonization but it is not clear if it decreases the risk of SSI.

Historically, chlorhexidine has been studied and used in orthopedic and cardiac implant surgeries. Research on the use of chlorhexidine for SSI prevention in cesarean sections is limited. This study intends to evaluate the effectiveness of use of both chlorhexidine gluconate (CHG) wipe and vaginal scrub in reducing SSI in patients undergoing cesarean section that have previously been laboring. Patients will be randomized to one of two groups: wash with both a pre-operative CHG cloth prior to surgery and chlorhexidine gluconate vaginal scrub in addition to standard preoperative scrub as compared to standard preoperative scrub alone.

DETAILED DESCRIPTION:
The study will be offered to women who are admitted to undergo labor at Mount Sinai Medical Center. The eligible women will be randomized to use of a 2% chlorhexidine gluconate (CHG) cloth with 4% chlorhexidine gluconate vaginal scrub (including standard preoperative care prior to cesarean section) or standard preoperative care. Participants will not be blinded to the arm in which they have been assigned.

Researchers will have access to all patients scheduled for delivery at Mount Sinai Medical Center. About 1800 deliveries by cesarean section occur each year at Mount Sinai. Of these, approximately 800 are cesarean sections after failed labor. Assuming a primary outcome rate of 20% in the control arm, a sample size of 329 in each group would give 80% power to detect a 40% reduction in surgical site infection between the active group and control. The aim is to recruit 400 patients per group (for a total of 800 patients) to account for patient drop out or non-compliance.

Sage Products, Inc will be providing the CHG cloths.

This study intends to show that simultaneous use of 2% CHG cloths and 4% CHG vaginal scrub prior to cesarean section will reduce the rate of SSI in women who have previously been laboring.

ELIGIBILITY:
Inclusion Criteria:

* Women at > 24 weeks gestation who are admitted in labor or admitted for induction of labor at Mount Sinai Hospital

Exclusion Criteria:

* Allergy to chlorhexidine
* Unplanned or emergency cesarean section
* Women at <24 weeks gestation
* Estimated fetal weight <500 grams
* Fetal face presentation regardless of gestational age.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 319 (Actual)
Dates: Start 2018-10-05 (Actual); Primary Completion 2021-02-11 (Actual); Study Completion 2021-02-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angela Bianco, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Background] Ahmed MR, Aref NK, Sayed Ahmed WA, Arain FR. Chlorhexidine vaginal wipes prior to elective cesarean section: does it reduce infectious morbidity? A randomized trial. J Matern Fetal Neonatal Med. 2017 Jun;30(12):1484-1487. doi: 10.1080/14767058.2016.1219996. Epub 2016 Sep 1. PMID 27583685
- [Background] Caissutti C, Saccone G, Zullo F, Quist-Nelson J, Felder L, Ciardulli A, Berghella V. Vaginal Cleansing Before Cesarean Delivery: A Systematic Review and Meta-analysis. Obstet Gynecol. 2017 Sep;130(3):527-538. doi: 10.1097/AOG.0000000000002167. PMID 28796683
- [Background] Culligan PJ, Kubik K, Murphy M, Blackwell L, Snyder J. A randomized trial that compared povidone iodine and chlorhexidine as antiseptics for vaginal hysterectomy. Am J Obstet Gynecol. 2005 Feb;192(2):422-5. doi: 10.1016/j.ajog.2004.08.010. PMID 15695981
- [Background] Darouiche RO, Wall MJ Jr, Itani KM, Otterson MF, Webb AL, Carrick MM, Miller HJ, Awad SS, Crosby CT, Mosier MC, Alsharif A, Berger DH. Chlorhexidine-Alcohol versus Povidone-Iodine for Surgical-Site Antisepsis. N Engl J Med. 2010 Jan 7;362(1):18-26. doi: 10.1056/NEJMoa0810988. PMID 20054046
- [Derived] Hadiati DR, Hakimi M, Nurdiati DS, Masuzawa Y, da Silva Lopes K, Ota E. Skin preparation for preventing infection following caesarean section. Cochrane Database Syst Rev. 2020 Jun 25;6(6):CD007462. doi: 10.1002/14651858.CD007462.pub5. PMID 32580252
- [Derived] Haas DM, Morgan S, Contreras K, Kimball S. Vaginal preparation with antiseptic solution before cesarean section for preventing postoperative infections. Cochrane Database Syst Rev. 2020 Apr 26;4(4):CD007892. doi: 10.1002/14651858.CD007892.pub7. PMID 32335895

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment and enrollment occurred between Oct 2018 and Feb 2021 at Mount Sinai Hospital's Labor and Delivery floor
Groups:
- Chlorhexidine Gluconate Vaginal Scrub and Cloth: Patients had a 2% chlorhexidine gluconate cloth applied to their abdomen as well as 4% chlorhexidine gluconate vaginal scrub applied as a vaginal cleanse in the operating room prior to cesarean section
  2% chlorhexidine gluconate cloth: applied to their abdomen
  4% Chlorhexidine gluconate vaginal scrub: applied as a vaginal cleanse in the operating room prior to cesarean section
- Standard Treatment: Patients who are not in the intervention arm received the standard of care prior to a cesarean section. In the operating room the patient will receive an abdominal cleanse with 2% Chloraprep solution (2% chlorhexidine gluconate) in addition to routine IV antibiotics.
  2% chlorhexidine gluconate cloth: applied to their abdomen
Period: Overall Study
Arm/Group | Chlorhexidine Gluconate Vaginal Scrub and Cloth | Standard Treatment
Started | 160 | 159
Completed | 152 | 150
Not Completed | 8 | 9
Not completed — Lost to Follow-up | 5 | 8
Not completed — Withdrawal by Subject | 1 | 0
Not completed — withdrawn due to vaginal delivery | 1 | 0
Not completed — Age < 18 | 1 | 0
Not completed — No Trial of Labor | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chlorhexidine Gluconate Vaginal Scrub and Cloth | Standard Treatment | Total
Number analyzed (Participants) | 160 | 159 | 319
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.01 (6.10) | 32.59 (5.43) | 32.30 (5.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 160 | 159 | 319
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 32 | 30 | 62
  Not Hispanic or Latino | 98 | 108 | 206
  Unknown or Not Reported | 30 | 21 | 51
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 15 | 16 | 31
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 25 | 28 | 53
  White | 64 | 67 | 131
  More than one race | 45 | 35 | 80
  Unknown or Not Reported | 11 | 12 | 23

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Surgical Site Infection
Description: Surgical site infection will be a composite of wound infection and postpartum endometritis. Endometritis is defined as postoperative fever of 100.4 °F or more occurring 24 hours after delivery associated with uterine tenderness and persistent foul-smelling lochia, requiring broad-spectrum intravenous antibiotic administration. Wound infection is defined as erythema or wound edge separation with purulent discharge involving the cesarean incision site that requires antibiotic therapy and wound care.
Time Frame: up to 6 weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Chlorhexidine Gluconate Vaginal Scrub and Cloth | Standard Treatment
Number analyzed (Participants) | 160 | 159
Participants | 12 | 22

2. Secondary Outcome: Number of Participants With Maternal Complications or Interventions
Time Frame: up to 6 weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Chlorhexidine Gluconate Vaginal Scrub and Cloth | Standard Treatment
Number analyzed (Participants) | 160 | 159
Participants | 7 | 1

3. Secondary Outcome: Number of Participants With Neonatal ICU Admissions
Description: Number of participants with newborn with neonatal ICU admissions
Time Frame: up to 6 weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Chlorhexidine Gluconate Vaginal Scrub and Cloth | Standard Treatment
Number analyzed (Participants) | 160 | 159
Participants | 30 | 36

4. Secondary Outcome: Maternal Length of Stay
Time Frame: up to 6 weeks postpartum
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Chlorhexidine Gluconate Vaginal Scrub and Cloth | Standard Treatment
Number analyzed (Participants) | 160 | 159
days | 2.98 (1.24) | 2.93 (0.78)

5. Secondary Outcome: Number of Participants With Readmissions
Time Frame: up to 6 weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Chlorhexidine Gluconate Vaginal Scrub and Cloth | Standard Treatment
Number analyzed (Participants) | 160 | 159
Participants | 6 | 2

6. Secondary Outcome: Estimated Blood Loss
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Chlorhexidine Gluconate Vaginal Scrub and Cloth | Standard Treatment
Number analyzed (Participants) | 160 | 159
mL | 671 (389) | 670 (391)

7. Secondary Outcome: Length of Time From Incision to Delivery
Time Frame: Day 1
Population: Data not collected
Arm/Group | Chlorhexidine Gluconate Vaginal Scrub and Cloth | Standard Treatment
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Length of Operation
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Chlorhexidine Gluconate Vaginal Scrub and Cloth | Standard Treatment
Number analyzed (Participants) | 160 | 159
Participants
  45-60 minutes | 46 | 46
  61-90 minutes | 87 | 96
  91+ minutes | 27 | 17

ADVERSE EVENTS:
Time Frame: up to 6 weeks postpartum
Arm/Group | Chlorhexidine Gluconate Vaginal Scrub and Cloth | Standard Treatment
All-Cause Mortality (participants affected / at risk) | 0/160 | 0/159
Serious Adverse Events (participants affected / at risk) | 0/160 | 0/159
Other Adverse Events (participants affected / at risk) | 0/160 | 0/159

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-11): https://cdn.clinicaltrials.gov/large-docs/47/NCT03423147/Prot_SAP_000.pdf